CLINICAL TRIAL: NCT05197439
Title: Effect of Dexmedetomidine on Postoperative Delirium in Elderly Patients With Parkinson's Disease Undergoing Deep Brain Stimulation: a Randomized Controlled Trial
Brief Title: Dexmedetomidine Prevents Postoperative Delirium After Deep Brain Stimulation in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20220106
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Dexmedetomidine; Postoperative Delirium; Deep Brain Stimulation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Active Comparator): Dexmedetomidine will be given at the beginning of the second step of DBS and last for 48 hours by electronic pump.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): The placebo group patients will be received 0.9% saline intraoperatively and postoperatively the same duration just like the DEX group would do.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Dexmedetomidine — The 4.8ug/kg dexmedetomidine will be diluted into 100ml and pump 2ml/h at the beginning of the second of DBS and last for 48 hours.
  Arms: DEX group
Drug: 0.9% saline — The 0.9% saline is administered with the same volume at the same speed as the other group.
  Arms: Placebo group

SUMMARY:
Postoperative delirium (POD) is a common complication, and the incidence of POD after deep brain stimulation(DBS) implementation ranges from 10% to 40%. Previous studies suggested that aging and existing non-motor symptom were independent risk factors for POD after supratentorial tumor resections. Therefore, patients undergoing DBS are high-risk populations for POD. A lot of trials show that dexmedetomidine might help to reduce the incidence of delirium in patients undergoing non-cardiac surgery. However, the impact of dexmedetomidine on POD for patients undergoing DBS was seldom reported. The purpose of this study was to investigate the effect of dexmedetomidine on POD in patients with Parkinson' Disease undergoing DBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease
* Exist non-motor symptoms
* Undergoing selective DBS.
* Age ≥60 years.
* Obtain written informed consent.

Exclusion Criteria:

* preoperative severe cognitive impairment (Montreal Cognitive Assessment, MoCA< 18)
* history of psychoactive
* allergic or intolerant to dexmedetomidine
* severe bradycardia (heart rate lower than 40 beats/min) or sick sinus syndrome, second-degree or third-degree atrioventricular block
* severe hepatic dysfunction (Child-Pugh class C)
* severe renal dysfunction requiring renal replacement therapy before the surgery
* medical records documented inability to communicate in the preoperative period due to language barrier or other situations.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium. | Postoperative 5 days
  Postoperative delirium is assessed by the combination of the Richmond Anxiety Scale (RASS) and the Confusion assessment method for intensive care unit (CAM-ICU) or the 3-minute diagnostic interview for CAM (3D-CAM) as applicable.

SECONDARY OUTCOMES:
The severity of postoperative delirium. | Postoperative 5 days
  The severity of postoperative delirium will be assessed by Delirium Rating Scale-Revised-98.
Postoperative pain | within 3 days after surgery.
  Postoperative pain will be assessed with Numerical Rating Scale (NRS). Postoperative analgesia will be recorded.
Quality of recovery. | First day after surgery
  Quality of recovery will be evaluated with 15-item quality of recovery questionnaire (QoR-15).
Quality of sleep | the second and the third day after surgery
  Quality of sleep will be evaluated with the Richards Campbell sleep questionnaire (RCSQ).
Cognitive function | before surgery and 5 days after surgery
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE) and the Montreal cognitive assessment-basic (MoCA-B).
Anxiety and depression | before surgery and 5 days after surgery
  Anxiety and depression will be evaluated using Generalized Anxiety Disorder-7 (GAD-7) and Patient Health Questionaire-9 items (PHQ -9).
Parkinson's disease related status | before surgery and 5 days after surgery
  Parkinson's disease related status will be evaluated by Movement Disorder Society-Sponsored Revision Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, MD,Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao J, Shen Z, Jin H, Ma T, Wang J, Li S, Zeng M, Liu X, Peng Y. Dexmedetomidine after deep brain stimulation for prevention of delirium in elderly patients with Parkinson's disease: protocol for a single-centre, randomised, double-blind, placebo-controlled trial in China. BMJ Open. 2023 Jul 11;13(7):e070185. doi: 10.1136/bmjopen-2022-070185. PMID 37433729